CLINICAL TRIAL: NCT01071538
Title: Buprenorphine for Late-Life Treatment Resistant Depression
Acronym: BUILD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Reckitt Benckiser LLC (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Jordan F. Karp, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUILD; KL2RR024154 (NIH)
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: Depressive Disorder, Major; Late-Life Depression; Geriatrics; Buprenorphine
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buprenorphine (Experimental): Older adults with treatment resistant depression will receive buprenorphine up to 1.6 mg/day for 8 weeks. Discontinuation of the buprenorphine will occur during weeks 9-12.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Sublingual buprenorphine 0.2 mg will be used for the first week. The dose will be increased by 0.2 mg/week based on safety and clinical response up to a maximal dose of 1.6 mg/day.

SUMMARY:
The goals of this pilot study are to gather data about the safety and clinical effect of low-dose buprenorphine in older adults with treatment resistant depression.

DETAILED DESCRIPTION:
We are recruiting 20 participants for this pilot study. Subjects are recruited from either:

1) An ongoing study of Late-Life Depression(MH083660; PI: Reynolds) who did not meet research response criteria; and 2) community-dwelling individuals, at least 50 years old, who have tried at least two FDA-approved antidepressant medications at therapeutic doses each for at least 6 weeks, and who are currently in an episode of major depression.

Overview of intervention: To guide future placebo-controlled work, at this preliminary stage of research we will collect data about both buprenorphine (BUP) 1) augmentation pharmacotherapy, and 2) monotherapy. Subjects recruited from the community will have the buprenorphine prescribed as augmentation to any currently prescribed antidepressant medication.

BUP 0.2 mg will be used for the first week. The first dose will be administered at the clinic under the supervision of the PI. Because peak plasma levels occur 60 minutes after ingestion, subjects will be re-assessed after 1 hour for safety. Participants will be seen weekly for eight weeks to assess progress and monitor intervention-emergent side effects. Dosing increases will be guided by antidepressant response (e.g., continued MADRS scores > 10 will trigger an increase dose of BUP) and our protocolized use of the Frequency, Intensity, and Burden of Side Effect Rating (FIBSER) Scale score. For example, a score of 5 to 7 on the FIBSER will trigger additional assessment of side effects and require justification for increasing the dose, while a score of > 7 will signal no increase in dose, although specific side effects should be reviewed in detail before a final determination, including review if the UKU Side Effects Rating Scale.

We will increase the dose by 0.2 mg/week up to 1.6 mg/day based on MADRS and FIBSER scores. Every time the dose is increased, the first ingestion of the higher dose will be monitored in the clinic as described above.

Subjects will participate in the project at the Late-Life Depression Clinic on the 7th Floor of Bellefield Tower. Subjects will complete paper and pencil and clinician-administered psychiatric assessments before receiving the first dose of buprenorphine and at all subsequent visits. After the first ingestion and all subsequent first ingestions of higher doses of BUP, subjects will remain in the clinic for 60 minutes after ingestion and be re-assessed for the emergence of side effects and have vital signs re-checked. The duration of the first visit will be approximately 2.5 hours. If subsequent visits require observed ingestion of buprenorphine, they will last about 1.75 hours. If subsequent visits do not require observed ingestion of buprenorphine, these visits will last 30-45 minutes.

Prior to the first ingestion, the first ingestion of subsequent higher doses, and at study end, subjects will complete a 15 minute battery of computerized neuropsychological tests assessing reaction time and attention. These tests will be repeated 60 minutes after the ingestion. Prior to the first ingestion and after discontinuation of the buprenorphine, memory will be assessed with the Hopkins Verbal Learning Test (HVLT). The HVLT takes about 10 minutes to complete.

The discontinuation phase will occur during weeks 9-12. To minimize the risk of withdrawal symptoms, we will discontinue the buprenorphine slowly by reducing the dose to 0.4 mg/day for 7 days, then 0.2 mg/day every other day for 7 days, and then stop the buprenorphine. We will see subjects weekly over these four weeks.

The final visit will occur at week 16. This will be a telephone check in of mood and functioning. This call will take about 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 50 years
* Major depressive disorder
* Non-responder to at least 2 FDA-approved antidepressants prescribed at a therapeutic dose, each for at least 6 weeks, or is a depression non-responder from an ongoing study of late-life depression at our research clinic.

Exclusion Criteria:

* Concomitant use of strong or moderate CYP3A4 inhibitor.
* Refusal to stop all opioids.
* Refusal to discontinue all alcohol.
* Refusal to discontinue benzodiazepines other than the equivalent of lorazepam 2 mg/day prescribed at a stable dose for at least the past 2 weeks.
* Hepatic impairment (AST/ALT > 1.5 times upper normal.
* Lung disease requiring supplemental oxygen.
* Estimated creatinine clearance <30 mL/min.
* Inability to provide informed consent.
* Depressive symptoms not severe enough (i.e., MADRS < 10) at the baseline assessment.
* Dementia.
* Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
* Abuse of or dependence on alcohol or other substances within the past 3 months.
* Meets criteria for history of abuse or dependence upon opioids.
* High risk for suicide.
* Contraindication to buprenorphine.
* Inability to communicate in English.
* Non-correctable clinically significant sensory impairment.
* Unstable medical illness.
* Subjects taking psychotropic medications that cannot be safely tapered and discontinued prior to study initiation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan F Karp, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinica, University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mague SD, Pliakas AM, Todtenkopf MS, Tomasiewicz HC, Zhang Y, Stevens WC Jr, Jones RM, Portoghese PS, Carlezon WA Jr. Antidepressant-like effects of kappa-opioid receptor antagonists in the forced swim test in rats. J Pharmacol Exp Ther. 2003 Apr;305(1):323-30. doi: 10.1124/jpet.102.046433. PMID 12649385
- [Background] Nyhuis PW, Gastpar M, Scherbaum N. Opiate treatment in depression refractory to antidepressants and electroconvulsive therapy. J Clin Psychopharmacol. 2008 Oct;28(5):593-5. doi: 10.1097/JCP.0b013e31818638a4. No abstract available. PMID 18794671
- [Background] Bodkin JA, Zornberg GL, Lukas SE, Cole JO. Buprenorphine treatment of refractory depression. J Clin Psychopharmacol. 1995 Feb;15(1):49-57. doi: 10.1097/00004714-199502000-00008. PMID 7714228
- [Background] Emrich HM, Vogt P, Herz A. Possible antidepressive effects of opioids: action of buprenorphine. Ann N Y Acad Sci. 1982;398:108-12. doi: 10.1111/j.1749-6632.1982.tb39483.x. No abstract available. PMID 6760767
- [Derived] Karp JF, Butters MA, Begley AE, Miller MD, Lenze EJ, Blumberger DM, Mulsant BH, Reynolds CF 3rd. Safety, tolerability, and clinical effect of low-dose buprenorphine for treatment-resistant depression in midlife and older adults. J Clin Psychiatry. 2014 Aug;75(8):e785-93. doi: 10.4088/JCP.13m08725. PMID 25191915
- See also: This link describes our other work with late-life depression at our NIH-funded research clinic in Pittsburgh, PA — http://www.ADAPTstudy.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: measure of depression severity theoretical scale range 0-60 Lower values represent better outcome
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine
Number analyzed (Participants) | 15
units on a scale | 9.5 (9.5)

2. Primary Outcome: Blood Pressure
Description: Blood Pressure- systolic and diastolic 140/90 or lower is considered normal and indicates a better outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Buprenorphine
Number analyzed (Participants) | 13
mm Hg
  systolic blood pressure | 122.5 (23.0)
  diastolic blood pressure | 70.5 (12.1)

3. Primary Outcome: UKU Side Effect Rating Scale
Description: measure of side effects 46 items with scores of 0,1,2,3 possible. Theoretical range 0-138 Lower scores indicate fewer side effects
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine
Number analyzed (Participants) | 13
units on a scale | 6.2 (3.5)

4. Secondary Outcome: Brief Symptom Inventory -- Anxiety Subscale
Description: measure of anxiety Lower numbers indicate better outcome Theoretical Range 0-2.4
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine
Number analyzed (Participants) | 13
units on a scale | 0.6 (0.8)

5. Secondary Outcome: Positive and Negative Affect Scale
Description: Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Score: Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine
Number analyzed (Participants) | 13
units on a scale
  Positive affect subscale | 29.4 (12.0)
  Negative affect subscale | 15.5 (6.7)

6. Secondary Outcome: Pain Numeric Rating Scale (20 Item)
Description: measure of average physical pain score range 0-20 Higher scores indicate worse outcome
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine
Number analyzed (Participants) | 13
units on a scale | 4.6 (5.2)

7. Primary Outcome: Heart Rate
Description: Heart Rate (Beats per minute) 60-100 beats per minute is considered normal lower heart rate represent healthier outcome
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Buprenorphine
Number analyzed (Participants) | 13
beats per minute | 72.7 (9.9)

ADVERSE EVENTS:
Arm/Group | Buprenorphine
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (N=15)
constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No